CLINICAL TRIAL: NCT02144311
Title: Benchmarking Intra-tumor Heterogeneity In Ovarian Cancer: Linking In-vivo Imaging Phenotypes With Histology And Genomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-061
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Ovarian Cancer
Keywords: MRI; FDG PET/CT; histologic heterogeneity; 14-061
MeSH Terms: conditions — Ovarian Neoplasms

ARMS (1):
- MRI with DW-MRI & DCE-MRI & FDG PET/CT (Experimental): Study participants will have 1 scan within the 7 days immediately preceding surgery (PET/CT as standard of care and MRI as a research exam). MRI and PET/CT scanning procedures will be identical to those used in routine clinical examinations of the abdomen and pelvis.
  Interventions: Procedure: PET/CT Scan; Procedure: MRI

INTERVENTIONS:
Procedure: PET/CT Scan
Procedure: MRI

SUMMARY:
The purpose of this research study is to learn if differences seen in scans before surgery match differences seen when looking at tumor samples with pathology and genetic tests. In this study we will use Magnetic Resonance Imaging [MRI] and Positron Emission Tomography [PET] scans. No direct clinical benefits will come from the results of this study.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age on the day of signing the informed consent.
* Histologically confirmed or suspected stage III or IV high-grade serous ovarian cancer.
* Scheduled to undergo primary debulking surgery.

Exclusion Criteria:

* Pregnant patients
* Patients who because of general medical or psychiatric condition, or physiologic status unrelated to the presence of ovarian cancer cannot give valid informed consent
* Patients who are unwilling or unable to undergo MRI including patients with contraindications to MRI such as the presence of cardiac pacemakers or non-compatible intracranial vascular clips, claustrophobia, inability to lie flat for the duration of the study etc.
* Patients with a metallic hip implant or any other metallic implant or device in the pelvis that might distort local magnetic field and compromise quality of MRI/
* Radiotherapy to the abdomen or pelvis within 6 months of the screening visit. Subjects with a current diagnosis of epithelial ovarian tumor of low malignant potential (borderline carcinomas) are not eligible
* Patients with synchronous primary endometrial cancer or a past history of endometrial cancer, unless all of the following conditions are met:
* Stage not greater than IB
* No more than superficial myometrial invasion
* No vascular or lymphatic invasion
* No poorly differentiated subtypes, including serous, clear cell, or other FIGO Grade 3 lesions.
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor are excluded. Patients who have received neoadjuvant chemotherapy prior to their initial debulking are excluded. Patients may have received prior adjuvant chemotherapy for breast cancer.
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, subjects with other invasive malignancies who had (or have) any evidence of the other cancer present within the last 3 years are excluded.
* Unresolved bowel obstruction.
* History or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with patient's participation for the full duration of the study.
* Absence of target lesions (> 2.0 cm) on staging CT
* Patients unlikely to be optimally debulked at surgery (tumor implants in difficult to reach places [i.e. falciform ligament or porta hepatis], suprarenal retroperitoneal lymphadenopathy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Genomic markers of spatial heterogeneity | 1 year
  by evaluating spatially explicit phenotypic clusters based on a combination of perfusion, diffusion and metabolic tumor profiles (maps) in both ovarian tumors and metastatic peritoneal/omental implants of patients with HGSOC undergoing primary debulking surgery (PDS).

SECONDARY OUTCOMES:
Histological and immunohistochemical features | 1 year
  The analyses involving the bioinformatic algorithms will be handled by the Bioinformatics Core. Previously validated bioinformatic algorithms (5, 13, 38) will be used to determine the clonal compositions of the imaging-based phenotypically distinct clusters of HGSOCs, and phylogenetic trees based on allelic frequencies of mutations and copy number aberrations of the primary ovarian tumor and matched metastatic implant will be constructed for each case

CONTACTS AND LOCATIONS:
Overall Officials: Hebert Vargas Alvarez, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/